CLINICAL TRIAL: NCT06309446
Title: Assessment of Wound Healing, Cooling Efficacy and Local Tolerability of a Wound Care Hydrogel With Intraindividual Comparison Using an Abrasive Wound Model in a Single-center, Randomized, Investigatorblind Clinical Investigation.
Brief Title: Assessment of Wound Healing, Cooling Efficacy and Local Tolerability of a Wound Care Hydrogel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 381001BS
Record Dates: First submitted 2024-02-28; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Wound
Keywords: Wound healing
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zoralan Wound (Experimental): At the beginning of the study, two small, superficial, abrasive wounds (approximately 1.2 cm in diameter) were induced on one volar forearm of each subject with a minimum distance of 5 cm between the wounds, using a sterile surgical hand brush.
  One wound is treated with the medical device by a study nurse and covered with standard semi-occlusive wound plaster (Hansaplast Sensitive wound plaster. Topical application of appoximately 0.2g per test field (approx. 1.2cm in diameter each) once daily during a 12-day treatment period (11 treatments).
  Interventions: Device: Zoralan Wound
- No treatment (No Intervention): At the beginning of the study, two small, superficial, abrasive wounds (approximately 1.2 cm in diameter) were induced on one volar forearm of each subject with a minimum distance of 5 cm between the wounds, using a sterile surgical hand brush.
  One wound is not treated but covered with standard semi-occlusive wound plaster (Hansaplast Sensitive wound plaster. Covering happens once daily during a 12-day treatment period (11 treatments).

INTERVENTIONS:
Device: Zoralan Wound — Topical application of approximately 0.2 g per test field (approx. 1.2 cm in diameter each) once daily during a 12-day treatment period (11 treatments).
  Other Names: Flamozil; Wound care hydrogel; X92001574
  Arms: Zoralan Wound

SUMMARY:
Test the wound healing properties of the product as well as the cooling effect and tolerability of a wound care gel.

DETAILED DESCRIPTION:
The primary goal of the study is to assess the wound healing properties in the test fields, based on the level of re-epithelialization, and to assess the cooling properties in the test fields, immediately after the first application of the Medical Device. The secondary objective was to assess the local tolerability of the test fields after inducing the wounds. The cosmetic outcome was assessed by the investigator and by the subject after 31 days using a visual analog scale (VAS) and by the subjects on day 12 by filling a questionnaire on product performance and times to 100% healing, over 75% healing respectively were derived from the re-epithelization score.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older;
* Healthy skin on the volar forearms;
* The physical examination of the skin must be without disease findings unless the investigator considers an abnormality to be irrelevant to the outcome of the clinical investigation;
* Female volunteers of childbearing potential must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices (IUDs), sexual abstinence or vasectomized partner;
* Urine pregnancy test negative for all females;
* Written informed consent obtained.

Exclusion Criteria:

* Acne, suntan, eczema, scars, excessive hair, acute skin infection or skin disease, hyper or hypopigmentation or tattoos in the test fields;
* Dark-skinned persons (Fitzpatrick skin types IV-VI);
* Pregnancy or planned pregnancy or nursing;
* Symptoms of a clinically significant illness that may influence the outcome of the investigation in the 4 weeks before baseline and during the clinical investigation;
* Participation in the treatment phase in another clinical investigation or clinical trial within the last 4 weeks prior to the baseline visit of this clinical investigation and during the conduct of this investigation;
* Known hypersensitivity or known allergic reactions to components of the MD or the protective standard wound plaster used;
* Treatment with systemic medications or medications acting locally in the test field areas which might counter or influence the investigation aim within 2 weeks before the baseline visit (e.g. antihistamines or glucocorticosteroids) and during the conduct of this investigation;
* Subjects who have taken any anticoagulant medication, within 3 weeks prior to Day 1, or platelet aggregation inhibitors within 10 days prior to Day 1 or with a history of hemophilia or any other illness influencing the subject's coagulation system.
* Subjects with diabetes mellitus or presence or history of psoriasis, atopic dermatitis, lichen ruber planus, impaired wound healing or keloid development;
* Contraindications according to the package leaflet/instructions of use (Hansaplast Sensitive);
* If in the opinion of the investigator or physician performing the initial examination the subject should not participate in the clinical investigation, e.g. due to probable noncompliance or inability to understand the investigation and adequately given informed consent;
* Subjects not willing to adhere to trial restrictions, amongst others sauna, solarium are not allowed during the clinical investigation;
* Close affiliation with the investigator (e.g. a close relative) or persons working at bioskin GmbH or subject is an employee of the sponsor;
* Subject with a disposition to develop hypertrophic scarring, keloids or wound healing disorders;
* Evidence of drug or alcohol abuse;
* Subject is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Wound healing efficacy (clinical) | Day 2, Day 6, Day 8, Day 10 & Day 12
  Clinical assessment of wound healing efficacy performed by investigator (6-point- reepithelialization score).
  0 = 0% healing
  1. = 1-25% re-epithelialization
  2. = 26-50% re-epithelialization
  3. = 51-75% re-epithelialization
  4. = over 75% but not complete re-epithelialization
  5. = 100% complete healing
Wound healing efficacy (global) | Day 2, Day 6, Day 8, Day 10 & Day 12
  Global assessment of wound healing efficacy performed by investigator (5-point score).
  0 = very good
  1. = good
  2. = acceptable
  3. = poor
  4. = very poor
Cooling properties | Day 1
  Subjective assessment of cooling properties performed by subject by completing a visual analogue scale on Day 1 immediately after application of the Medical Device (MD).The cooling effect in the two test fields will be assessed by the subject by means of a visual analogue scale (VAS) of 100 mm length, ranging from 0 (no cooling) to 100 (extremely cooling) on Day 1, 20 ±5 seconds after application of the MD (but prior to application of the protective wound plaster).

SECONDARY OUTCOMES:
Local tolerability (clinical) | Day 2, Day 6, Day 8, Day 10 & Day 12
  Clinical assessment of local tolerability performed by investigator (5-point-erythemascore).
  0 = no reaction
  1. = slight uniform or spotty erythema or slight diffuse, partial or follicular erythema
  2. = clear, sharply demarcated erythema
  3. = severe erythema with infiltrate
  4. = severe erythema with infiltrate and/or epidermal defect (blisters, blebs, erosions)
Local tolerability (global) | Day 2, Day 6, Day 8, Day 10 & Day 12
  Global assessment of local tolerability performed by subject and investigator (5-point score). 0 = very good
  1. = good
  2. = acceptable
  3. = poor
  4. = very poor
Signs of infection | Day 2, Day 6, Day 8, Day 10 & Day 12
  Assessment of signs of infection, considering the following parameters: erythema, pain, malodor, delayed wound healing, excessive exudate, and heat, by investigator (closed question: YES/NO).
Time until 100% healing | Day 2, Day 6, Day 8, Day 10 & Day 12
  Time until 100% healing, defined as first day after wound induction with reepithelialization score of 5 (5 = 100% complete healing).
Time until 75% healing | Day 2, Day 6, Day 8, Day 10 & Day 12
  Time until over 75% healing, defined as first day after wound induction with reepithelialization score of 4 or 5 (4 = over 75% but not complete re-epithelialization; 5 = 100% complete healing).
Presence of crusts | Day 2, Day 6, Day 8, Day 10 & Day 12
  Presence of crusts (Yes/No)
Questionnaire on product performance | Day 12
  Questionnaire on product performance (filled by subjects) on Day 12 (12 closed questions)
Cosmetic outcome/acceptance | Day 31
  The cosmetic outcome/acceptance will be assessed by the investigator and the subject by means of a visual analogue scale (VAS) of 100 mm length, ranging from 0 (poor) to 10 (excellent) on Day 31±2 for each of the two test fields.
Photographic documentation of the wound - visual of the wound to support previous outcomes. | Day 1, Day 4, Day 6, Day 8, Day 10, Day 12 & Day 31
  High-quality photographic documentation of the test sites on Days 1, 4, 6, 8, 10, 12 and 31 sufficient time (not earlier than 30 minutes but not later than 60 minutes) after removal of patches and product residues for any removal related erythema to subside.

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Siemetzki, M.D., Principal Investigator — Bioskin GmbH
Locations (1):
- Bioskin GmbH, Hamburg, Germany